CLINICAL TRIAL: NCT06113107
Title: Impact of Modifications to the Rendering of the Antibiogram on the Prescriptions of Meropenem in Pseudomonas Bacteremia
Acronym: Mero-Pyo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8786
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Pseudomonas
Keywords: Pseudomonas; Meropenem; Microbial susceptibility testing; EUCAST breakpoint; Antibiotic stewardship
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Modification of the rendering of the antibiogram at the Strasbourg University Hospital in November 2019 with the appearance of the concept of "standard dose" or "high dose" sensitivity.

This modification seems to have favored an inappropriate overprescription of Meropenem (the only antibiotic made "at standard dose") in Pseudomonas infections sensitive to other beta-lactams.

In June 2021, it was therefore decided to mask sensitivity to carbapenems by default in the rendering of Pseudomonas antibiograms when the strain was sensitive to a narrower spectrum beta-lactam ("restricted" antibiogram).

The aim of this study is to evaluate the impact of these changes in the antibiogram on antibiotic prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject with a positive blood culture result for Pseudomonas spp identified in the microbiology laboratory of Strasbourg University Hospital during the period from June 1, 2018 to November 30, 2022
* Subject not opposing the reuse of their data for the purposes of this research.

Exclusion Criteria:

* Subject having expressed opposition to participating in the study,
* Pseudomonas spp strain resistant to all first-line beta-lactams (Piperacillin-Tazobactam, Ceftazidime, Céfepime and Aztreonam).
* Pseudomonas spp strain resistant to Meropenem.
* Lack of information on the antibiotic treatment undertaken.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) with a positive blood culture result for Pseudomonas spp identified in the microbiology laboratory of Strasbourg University Hospital during the period from June 1, 2018 to November 30, 2022
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of Meropenem prescriptions in Pseudomonas spp bacteraemia susceptible to narrow-spectrum betalactams | Files analysed retrospectively from June 1, 2018 to November 30, 2022 will be examined
  This study is retrospective, the analysis focuses on the medical records of patients treated at the Strasbourg University Hospital between June 1, 2018 and November 30, 2022.

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France